CLINICAL TRIAL: NCT04355117
Title: A Multicenter, Open-label Trial to Evaluate the Safety of TEV-48125 When Subcutaneously Self-administered in Migraine Patients at the Trial Site and at Home
Brief Title: A Safety Evaluation Trial of TEV-48125 Self-administered in Migraine Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 406-102-00005
Record Dates: First submitted 2020-03-19; First posted 2020-04-21 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment: TEV-48125 (Experimental)
  Interventions: Drug: Each subject will subcutaneously self-administer TEV 48125 at 225 mg/1.5 mL (150 mg/mL) once monthly for a total of 2 doses.

INTERVENTIONS:
Drug: Each subject will subcutaneously self-administer TEV 48125 at 225 mg/1.5 mL (150 mg/mL) once monthly for a total of 2 doses. — Each subject will subcutaneously self-administer TEV 48125 at 225 mg/1.5 mL (150 mg/mL) once monthly for a total of 2 doses.

SUMMARY:
This trial assesses the safety of TEV-48125 when subcutaneously self-administered in Japanese migraine patients using an autoinjector (AI) at home. Each subject will subcutaneously self-administer TEV 48125 at 225 mg/1.5 mL (150 mg/mL) once monthly for a total of 2 doses. The first dose will be self-administered at the trial site under the supervision of the investigator and the second dose will be self-administered at home.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of migraine (according to the ICHD-3 criteria) diagnosis for ≥12 months prior to giving informed consent.
* Patient fulfills any of the migraine criteria(according to the ICHD-3 criteria) on ≥4 days in baseline information collected during the 28-day screening period

Exclusion Criteria:

* History of hypersensitivity reactions to injected proteins, including monoclonal antibodies
* Prior exposure to a monoclonal antibody targeting (CGRP) pathway meeting the following conditions:

  * Less than 5 months has passed since the final administration of AMG334, ALD304, or LY2951742.
  * Less than 1 year has passed since the final administration of TEV-48125

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Sendai Zutsu No-Shinkei Clinic, Sendai, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: TEV-48125: Each subject subcutaneously self-administered TEV-48125 at 225 mg/1.5 mL (150 mg/mL) using an autoinjector (AI) once monthly for a total of 2 doses. The first dose was self-administered at the trial site under the supervision of the investigator (Baseline) and the second dose was self-administered at home (Visit 3).
Period: Overall Study
Arm/Group | Treatment: TEV-48125
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: TEV-48125
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 71
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Treatment-emergent Adverse Event (TEAE)
Description: * TEAEs were defined as AEs that started after the start of investigational medicinal product (IMP) treatment; or if the event was continuous from baseline and was worsening after the start of IMP treatment.
  * The number of subjects with TEAEs were provided by self-administration at the trial site and by self-administration at home.
    1. For TEAEs following self-administration at the trial site, TEAEs that occurred after self-administration at the trial site (Baseline) but before self-administration at home (Visit 3) were tabulated.
    2. For TEAEs following self-administration at home, TEAEs that occurred after self-administration at home but before the end of the trial were tabulated.
Time Frame: [1] Baseline (Day 1) to Day 28, [2] Visit 3 (Day 29) up to end of treatment (Day 57)
Population: Safety Set: subjects who have received at least 1 dose of the IMP
Measure: Count of Participants; unit: Participants
Groups:
- Self-administration at Trial Site: Each subject subcutaneously self-administered TEV-48125 at 225 mg/1.5 mL (150 mg/mL) using an autoinjector (AI) once monthly at the trial site under the supervision of the investigator (Baseline).
- Self-administration at Home: Each subject subcutaneously self-administered TEV-48125 at 225 mg/1.5 mL (150 mg/mL) using an autoinjector (AI) once monthly at home (Visit 3).
Arm/Group | Self-administration at Trial Site | Self-administration at Home
Number analyzed (Participants) | 71 | 71
Participants | 18 | 26

2. Secondary Outcome: Execution Status of Self-administration - Amount of Drug Solution Remaining in the AI
Description: Following self-administration at the trial site and at home, the AI was checked to see whether or not all of the drug solution had been injected and the appropriate description of the amount of drug solution remaining in the AI was recorded based on th following 5-point scale (0 to 4) measure.
  * 0: All drug solution has been injected
  * 1: Approximately 1/4 of the drug solution remaining
  * 2: Approximately 1/2 of the drug solution remaining
  * 3: Approximately 3/4 of the drug solution remaining
  * 4: Almost all of the drug solution remaining
Time Frame: Baseline (Day 1) and Visit 3 (Day 29)
Population: Safety Set: subjects who have received at least 1 dose of the IMP
Measure: Count of Participants; unit: Participants
Arm/Group | Self-administration at Trial Site | Self-administration at Home
Number analyzed (Participants) | 71 | 71
Participants
  Reported as 0 | 71 | 70
  Reported as 1 | 0 | 1
  Reported as 2 | 0 | 0
  Reported as 3 | 0 | 0
  Reported as 4 | 0 | 0

3. Secondary Outcome: Execution Status of Self-administration - Leakage of Drug Solution on the Skin
Description: Following self-administration at the trial site and at home, the injection site was observed for any leakage of drug solution on the skin was recorded based on the following 5-point scale (0 to 4) measure. Criteria 0, 1, and 2 on the 5-point scale measure were deemed to represent a successful self-injection.
  * 0: No sign of drug solution on the skin
  * 1: Slight wetness on the skin (mist)
  * 2: Approx. 1/5 (0.3 mL) of the drug solution observed on the skin (most of the drug solution subcutaneously administered)
  * 3: Approx. 1/2 (0.75 mL) of the drug solution observed on the skin (ie, approx. 1/2 of drug solution subcutaneously administered)
  * 4: Almost all of the drug solution observed on the skin (ie, little or no drug solution subcutaneously administered)
Time Frame: Baseline (Day 1) and Visit 3 (Day 29)
Population: Safety Set: subjects who have received at least 1 dose of the IMP
Measure: Count of Participants; unit: Participants
Arm/Group | Self-administration at Trial Site | Self-administration at Home
Number analyzed (Participants) | 71 | 71
Participants
  Reported as 0 | 58 | 48
  Reported as 1 | 12 | 20
  Reported as 2 | 1 | 3
  Reported as 3 | 0 | 0
  Reported as 4 | 0 | 0

4. Secondary Outcome: Subject Compliance With the Self-administration Procedure
Description: Subject compliance with the self-administration procedure was evaluated based on information recorded on a checklist.
  Compliance with each of the procedures during IMP preparation, injection administration, and after injection was verified by checking the "Yes" or "No" responses marked for each item on the checklist. Based on this checklist, the investigator judged adherence to self-administration procedure.
Time Frame: Baseline (Day 1) and Visit 3 (Day 29)
Population: Safety Set: subjects who have received at least 1 dose of the IMP
Measure: Count of Participants; unit: Participants
Arm/Group | Self-administration at Trial Site | Self-administration at Home
Number analyzed (Participants) | 71 | 71
Participants
  Reported as "Yes" | 71 | 70
  Reported as "No" | 0 | 1

5. Secondary Outcome: Number of Deficiencies With the AI Device
Description: A deficiency with the AI device (AI device deficiency) is defined as any defect in the quality, safety, or performance of the device, such as mechanical breakage and malfunction, no matter whether it is caused by design, manufacture, dispensing, storage,or use.
Time Frame: Baseline (Day 1) and Visit 3 (Day 29)
Population: Safety Set: subjects who have received at least 1 dose of the IMP
Measure: Number; unit: deficiencies with the AI device
Arm/Group | Treatment: TEV-48125
Number analyzed (Participants) | 71
deficiencies with the AI device | 1

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to end of treatment (Day 57)
Description: Safety Set: subjects who have received at least 1 dose of the IMP
Arm/Group | Treatment: TEV-48125
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 33/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: TEV-48125 (N=71)
Lymphadenitis (Blood and lymphatic system disorders) | 1
Glaucomatocyclitic crises (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Injection site erythema (General disorders) | 18
Injection site haemorrhage (General disorders) | 3
Injection site induration (General disorders) | 11
Injection site pain (General disorders) | 6
Injection site pruritus (General disorders) | 4
Injection site swelling (General disorders) | 1
Injection site warmth (General disorders) | 1
Pyrexia (General disorders) | 2
Gallbladder polyp (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Nasopharyngitis (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Heat stroke (Injury, poisoning and procedural complications) | 1
Liver function test abnormal (Investigations) | 1
Liver function test increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT04355117/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04355117/SAP_001.pdf